





# A Comparison of innate immune responses induced by allergy immunotherapy with different adjuvants

The original Patient Info was composed in German. This document is an English translation (by google translate) thereof for the purpose of registering the trial on <a href="https://www.clincaltrials.gov">www.clincaltrials.gov</a>

This research project is organised by:

- Prof. Dr. sc. nat. Pål Johansen, Department of Dermatology, University Hospital Zurich, Gloriastrasse 31, 8091 Zurich, Switzerland
- Prof Dr. med. Ludger Klimek, Centre for Rhinology and Allergology, Wiesbaden, An den Quellen 10, 65183 Wiesbaden, Germany

Dear madam, dear sir,

We would like to ask you if you want to participate in a research project. Below you will find the planned research project:

# **Detailed information**

# 1. Project goal

We want to use this project to investigate whether immune reactions can be detected in the first few days after allergen immunotherapy (AIT) in blood. A blood sample should be taken before their appointment with the allergist and 1, 7 and 49 days later. This would allow us to test the immune reactions in the laboratory.

#### 2. Selection of participants

All persons suffering from and / or being treated for an allergic disease may participate. In addition, you must be older than 18 years.

# 3. General information about the project

It is a research project carried out at the University Hospital Zurich (CH) in cooperation with the Centre for Rhinology and Allergology, Wiesbaden (DE). The project will involve 24 patients (16 in Zurich and 8 in Wiesbaden) with rhino-conjunctivitis due to sensitization to grass pollen or birch pollen and who have scheduled for allergen immunotherapy in Zurich or Wiesbaden. Before immunotherapy and one day and seven days later, a blood sample will be collected as part of the research project. In laboratory studies, blood is analysed for inflammatory cells (e.g., leukocytes) and molecules (e.g., enzymes, cytokines, and antibodies). The aim is to test how the various immunotherapeutic adjuvants (immunoreaction enhancers) influence the measured inflammatory responses. The

research project is carried out in accordance with the legislation in forces in Switzerland and Germany. The responsible ethics committees has examined and approved this project.

#### 4. Procedures

If you give consent to participate in this project, you will be briefed by an investigator. If you meet the requirements for participating in the project, a blood sample will be taken shortly before your first immunotherapy session (first allergen injection). You will then be asked by the examiner to come back to the clinic one day, 7 days and approximately 49 (± 3) days later for further blood samples. The last blood sample is likely to coincide with the last immunotherapy session (second allergen injection). Approximately 61 millilitres (ml) of blood are taken: 17 ml each on days 0, 1 and 7, and 10 ml on day 49. At each session, you will have to answer a questionnaire together with the investigator. Filling out the questionnaire will take about 5 minutes at each session. After the last blood sample you will be discharged from the study

#### 5. Benefits

You will not personally benefit from participating in the project. Many research findings are not relevant for the individual patients. However, your participation in this project could help physicians and researchers to gain new insights into allergen-specific immunotherapy and the mechanisms of action of such treatment.

#### 6. Rights

Your participation in this study is voluntary. If you do not want to join or later withdraw your participation, you do not have to justify this. Your medical treatment / care is guaranteed regardless of your decision. You are always welcome to ask questions about participation and the project. Please contact the person mentioned at the end of this information.

#### 7. Duties

As a participant it is necessary that you (i) adhere to the necessary requirements and requirements by the project management, and (ii) appear on time for scheduled visits.

#### 8. Risks

When participating in the project, you are exposed to only minor risks. Blood collection may cause bruising and, in very rare cases, infection.

# 9. Results

The investigator will inform you during the seven-day research project about any new findings that may affect the benefit or your safety and thus your consent to participate. You will be informed of any incidental findings that may help prevent, detect or treat existing or future illnesses. As no drug or surgical treatment will be provided for this research study, only blood sampling, no results will be available during the seven-day research project. The results of the analysis will be available only after their release from the study. If you do not want to be informed, please talk to your investigator.

# 10. Confidentiality of data and samples

Your personal and medical data will be collected for this project. Very few professionals will see your unencrypted data, solely to fulfil project tasks. When collecting data for study purposes, the data is encrypted. Encryption means that any reference data that you could identify (name, date of birth) is deleted and replaced with a key. The key list always stays in

the institution (University Hospital Zurich or Allergy Centre Wiesbaden). Therefore, those people who do not know the key cannot draw any conclusions about you. For a publication, the summarized data is therefore not traceable to you as an individual. Her name never appears on the Internet or a publication. Sometimes there is a requirement for a magazine to publish that individual data (so-called raw data) must be transmitted. If individual data needs to be transmitted, then the data is always encrypted and therefore not traceable back to you as a person. All persons who have access to your data as part of the project are subject to secrecy. The requirements of data protection are complied with and you as a participating person have the right to access your data at any time.

When data or samples are stored on site, it is a database or biobank for research purposes.

Sample shipments to other research institutions in Switzerland or abroad are not planned. Should the data and samples be forwarded for further project-specific examination, they will be encrypted first and then sent. Only the leader of this project has access to this encryption. Responsible for compliance with national and international data protection guidelines is project management, which ensures equivalent data protection abroad.

This project may be reviewed by the responsible ethics committee or by the institution that initiated the project. The project manager may need to disclose your personal and medical data for such controls.

It is possible that your doctor will be contacted to provide information about your state of health.

#### 11. Regulatory insight into the study

The project Management will be given direct access to and access to the subject's original medical records upon request by the Ethics Committee or other health or regulatory authorities to review project procedures or data. This access is granted without violating their confidentiality

#### 12. Withdrawal of consent

Participation in this research project is voluntary. You can cancel your participation at any time and withdraw from the project, if you so desire. The data and samples collected so far are still being evaluated in encrypted form, because otherwise the whole project loses its value.

It is not possible to anonymize your data and samples upon withdrawal, i.e., the data and samples remain encrypted. Please check if you agree before joining the project.

#### 13. Compensation

If you participate in this project, you will not receive any compensation. If they have travel related to the study, they will be compensated by the project management.

#### 14. Liability

- A) Zurich: If you suffer any damage to health as a result of the study, the University Hospital Zurich ("Insurance for clinical trials and non-clinical trials", *Zurich Versicherung*, Insurance number 14.970.888)
- B) Wiesbaden: For patients who visit the AZW, the local patient insurance applies in the event of damage to health, as approved by Prof. Klimek of the Mannheim Ethics Committee.

# 15. Project financing

The project is funded by research funds from the University of Zurich.

# 16. Contact persons

For any uncertainty, fears or emergencies that arise during or after the project, you may contact one of these contacts at any time.

# **University Hospital Zurich:**

Prof. Dr. sc. nat. Pål Johansen (PI Zurich)

Email pal.johansen@usz.ch

Tel +41 (0)44 255 8616

Dr. med. Deborah Leuthard (Investigator)

Email deborah.leuthard@usz.ch

Tel +41 (0)43 253 0568

Dr. med. Sara Micaletto (Allergologist)

Email sara.micaletto@usz.ch

Tel +41 (0)43 253 7630

Dr. med Eugen Bersuch (Allergologist)

Email: eugen.bersuch@usz.ch

Tel +41 (0)43 253 8580

Frau Elvira Schmid (Head nurse, allergy unit)

Email elvira.schmid@usz.ch

Tel +41 (0)44 255 2441

Emergency USZ: Tel +41 (0)44 255 11 11

# Centre for Rhinology and Allergology, Wiesbaden:

Prof. Dr. med. Ludger Klimek (PI Wiesbaden) Email: ludger.klimek@allergiezentrum.org

Tel: +49 (0)611 308 608-0

Dr. med. Annette Sperl (Allergologist)
Email: <a href="mailto:annette.sperl@allergiezentrum.org">annette.sperl@allergiezentrum.org</a>

Tel: +49 (0)611 308 608-0

Cand. med. Alina Müller (Investigator)

Email: <u>alina.mueller@usz.ch</u> Tel: +41 (0)76 391 18 35

Dr. Ingrid Casper (Study coordinator)

Email ingrid.casper@allergiezentrum.org

Tel +49 (0)611 308 608-257







# Written patient consent to participate in a research study

- Please read this form carefully.
- Please ask if you do not understand or want to know something

# BASEC-Number (swissethics): 2019-01233

# Study code USZ-AZW\_MCT001

**Study name** A Comparison of innate immune responses induced by allergy immunotherapy with different adjuvants

**Sponsor** Dept. Dermatology, University Hospital Zurich & University of Zurich, Gloriastrasse 31, 8091 Zürich, Switzerland

**Study location** University Hospital Zurich (CH) and Centre for Rhinology and Allergology, Wiesbaden (DE)

**Principle investigators** Prof. Dr. sc. nat. Pål Johansen (Zurich), Prof. Dr. med. Ludger Klimek (Wiesbaden)

**Investigators** Dr. med. Deborah Leuthard (Zurich) und Dr. med. Annette Sperl (Wiesbaden), med. pract. Alina Müller (Zurich and Wiesbaden)

#### **Patient**

Name

Date of birth

Gender

female / male

- I have been informed verbally and in writing by the undersigned physician about the
  objectives and course of the USZ-AZW\_MCT001 study, the expected effects, possible
  benefits and disadvantages, and any risks.
- I have read and understood the written patient information of August 9, 2019 for the study mentioned above. My questions related to participation in this study have been satisfactorily answered to me. I can keep the written patient information and receive a copy of my written informed consent.
- I had sufficient time to make my decision.
- I am aware that an insurance covers damages if they occur in the study.
- I know that my data and samples can only be passed on in encrypted form within the framework of this study
- I agree that the investigators, the authorities and the Cantonal Ethics Commission may inspect my original data for checking and control purposes, but with strict confidentiality.

- I volunteer to participate in this study. I can revoke my consent to participate at any time and without stating reasons, without incurring any disadvantages in the further medical care. In that case, for my own safety, I will be examined medically.
- I am aware that the requirements and limitations stated in the patient information must be adhered to during the study. In the interest of my health, the investigator can always exclude me from the study.

| Place and date | Patient's signature |
|---|---|
| Confirmation backs investigation | |
| <b>Confirmation by the investigator:</b> I hereby certify that I have explained to this patient the nature, significance and scope of the study. I assure you to fulfil all obligations related to this study. If, at any time during the study, I am experiencing any issues that may affect the patient's willingness to participate in the study, I will promptly inform him / her. | |
| Place and date | Investigator's signature |